CLINICAL TRIAL: NCT05811117
Title: Multicenter Study Using Imaging Mass Cytometry to Analyze the Impact of ICANS on Microglia
Brief Title: Multicenter Study Using IMC to Analyze the Impact of ICANS on Microglia
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director Division of Tumor Immunology, University of Freiburg
Other Study IDs: UKLFR02022021
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: ICANS, Grade Unspecified; CAR T-Cell-Related Encephalopathy Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: There will be no intervention as we will study patients that undergo autopsy after CAR T cell infusion. — We will study patients that undergo autopsy after CAR T cell infusion.

SUMMARY:
Immunotherapy with chimeric antigen receptor (CAR) T cell therapy can cause immune effector cell-associated neurotoxicity syndrome (ICANS). However, the molecular mechanisms leading to ICANS are not well understood. In this study, the investigators plan to examine the role of microglia as the primary parenchymal immune cells of the central nervous system (CNS) during ICANS in human samples. The samples will be analyzed using imaging-mass-cytometry-based analysis (IMC). Single-cell data will be obtained through machine learning supervised segmentation of IMC data. Single-cell marker expression in all cells and in microglia (Iba1+ cells) will be analyzed in patients with ICANS.

DETAILED DESCRIPTION:
Immunotherapy with chimeric antigen receptor (CAR) T cell therapy can cause immune effector cell-associated neurotoxicity syndrome (ICANS).

Previous studies have shown a role for IL-1beta and IL-6 in xenograft mouse models.

However, the molecular mechanisms leading to ICANS are not well understood. In this study, the investigators plan to examine the role of microglia as the primary parenchymal immune cells of the central nervous system (CNS) during ICANS in human samples. The samples will be analyzed using imaging-mass-cytometry-based analysis (IMC). Single-cell data will be obtained through machine learning supervised segmentation of IMC data. Single-cell marker expression in all cells and in microglia (Iba1+ cells) will be analyzed in patients with ICANS. The participants are patients treated with chimeric antigen receptor (CAR) T cell therapy. The patients will received TSPO-PET imaging if available and if an autopsy is performed underroutine conditions tissue is collected for IMC based analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients that had developed ICANS
* CAR T cell infusion for lymphoid malignancy (NHL or ALL)

Exclusion Criteria:

* Lack of consent of patient or legal guardian

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that had developed ICANS after CAR T cell infusion will be analyzed.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
HLA-DRA and HLA-DR on Iba1+ cells | 2 years
  We will study HLA-DRA and HLA-DR on Iba1+ cells
Clusters of activated microglia and macrophages will be studied in patients with ICANS | 2 years
  Clusters of activated microglia and macrophages will be studied in patients with ICANS

CONTACTS AND LOCATIONS:
Locations (1):
- Freiburg University Medical Center, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zeiser R, Polverelli N, Ram R, Hashmi SK, Chakraverty R, Middeke JM, Musso M, Giebel S, Uzay A, Langmuir P, Hollaender N, Gowda M, Stefanelli T, Lee SJ, Teshima T, Locatelli F; REACH3 Investigators. Ruxolitinib for Glucocorticoid-Refractory Chronic Graft-versus-Host Disease. N Engl J Med. 2021 Jul 15;385(3):228-238. doi: 10.1056/NEJMoa2033122. PMID 34260836